CLINICAL TRIAL: NCT03066479
Title: Comparing Fitbit® Quality of Measured Sleep to Sleep Measured by Polysomnography in the Sleep Lab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vidya Raman (Other)
Responsible Party: Sponsor-Investigator, Vidya Raman, Clinical Associate Professor of Anesthesiology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB15-00331
Record Dates: First submitted 2017-02-16; First posted 2017-02-28 (Actual); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fitbit (Experimental): Patients will wear a Fitbit bracelet during their sleep study.
  Interventions: Device: Fitbit; Other: OSA questionnaire; Diagnostic Test: Polysomnography

INTERVENTIONS:
Device: Fitbit — Wearable activity & sleep tracker.
Other: OSA questionnaire — Parents will complete a questionnaire assessing the potential symptoms their child is experiencing that are related to obstructive sleep apnea (OSA).
Diagnostic Test: Polysomnography — All participants will be undergoing a sleep study as part of their clinical care.
  Other Names: Sleep study

SUMMARY:
This study is to evaluate a commercial tool on the market (Fitbit®) that also quantifies sleep. No one has studied how pediatric patients perform with it and how accurate it is in measuring their quality of sleep. This study will use the obstructive sleep apnea (OSA) questionnaire completed by parents and Fitbit® together and evaluate how they perform against the polysomnography (PSG).

ELIGIBILITY:
Inclusion Criteria:

* Patients who consent/assent to wearing Fitbit® band over wrist overnight during sleep study and parents who consent to answering questionnaire.

Exclusion Criteria:

* None

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08-04 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Total sleep time | At the end of the sleep study - average 6 hrs.
  Compare the sleep times recorded on the Fitbit vs the sleep study.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No